CLINICAL TRIAL: NCT01438411
Title: An Open Label, Single Center, Nonrandomized Continuation Study of Cholic Acid Capsules to Treat Subjects With Inborn Errors of Bile Acid Synthesis
Brief Title: Open Label, Continuation Study of Cholic Acid in Subjects With Inborn Errors of Bile Acid Synthesis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mirum Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAC-002-01
Record Dates: First submitted 2011-09-20; First posted 2011-09-22 (Estimated); Results first posted 2020-08-21 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Bile Acid Synthesis Defect
Keywords: Cholic Acid; Inborn Error; Bile Acid Metabolism; Inborn Error of Bile Acid Synthesis
MeSH Terms: interventions — Cholic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cholic Acid (Other): Active drug
  Interventions: Drug: Cholic Acid

INTERVENTIONS:
Drug: Cholic Acid — 10-15 mg/kg body weight/day supplied in 50 or 250 mg Cholic Acid Capsules
  Other Names: Cholic; Cholic Acid Capsules

SUMMARY:
The primary purpose of the study is to evaluate the therapeutic efficacy and safety of cholic acid in subjects with identified inborn errors of bile acid synthesis.

DETAILED DESCRIPTION:
This is a Phase 3, open-label, single center, nonrandomized study. This continuation protocol will consist of eligible subjects who have previously received cholic acid through the Cincinnati Children's Hospital Medical Center (CCHMC) Compassionate Use (91-10-10), CAC-001-01 study protocols and newly diagnosed subjects.

New subjects will be infants, children, adolescents identified from urine samples obtained from the clinical services of programs across the U.S., Canada, South America, Europe, and Asia. Subject or their legal representative will receive information regarding the study, and the principle investigator (PI) or designee will obtain informed consent. Serum and urine samples will be collected and sent to CCHMC to measure complete bile acid profile analysis. Clinical records including medical history, physical exams, vital signs, and laboratory assessments performed as standard of care will be reviewed to ensure subject eligibility and determine baseline values.

Subjects who have participated in Protocols conducted under IND 45,470 will be consented to continue to receive cholic acid capsules under this continuation protocol. Subjects will serve as their own controls and no placebo will be utilized.

ELIGIBILITY:
Inclusion Criteria:

Subjects who received cholic acid through CCHMC protocols 91-10-10 or CAC-002-01 and meet the following criteria are eligible for study participation.

1. The subject and/or parent/legal guardian must have provided informed consent prior to study start.
2. The subject must have a diagnosis of an inborn error of bile acid synthesis.
3. The subject must be willing and able to comply with all study assessments and procedures.
4. Subjects with other organ dysfunction will not be excluded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2010-01; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James E Heubi, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Kenneth Setchell, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Heubi JE, Setchell KDR. Open-label Phase 3 Continuation Study of Cholic Acid in Patients With Inborn Errors of Bile Acid Synthesis. J Pediatr Gastroenterol Nutr. 2020 Apr;70(4):423-429. doi: 10.1097/MPG.0000000000002618. PMID 31899729

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study included subjects with inborn errors of bile acid metabolism who had previously participated in studies CAC-91-10-10 or CAC-001-01 as well as newly diagnosed subjects.
  Data were collected from 1 Jan 2010 through study completion on 31 Jul 2016. Note that treatment with cholic acid continues throughout a subject's lifetime.
Pre-assignment Details: Of 53 subjects, 31 subjects rolled over from studies CAC-91-10-10 and/or CAC-001-01, while 22 patients were treatment-naive, i.e. received their first dose of cholic acid during study CAC-002-01.
Groups:
- Cholic Acid: Cholic acid capsules, each containing 50 mg or 250 mg of cholic acid to be administered orally at a daily dose of 10-15 mg/kg body weight
Period: Overall Study
Arm/Group | Cholic Acid
Started | 53
Completed | 40
Not Completed | 13
Not completed — Adverse Event | 8
Not completed — Lost to Follow-up | 1
Not completed — Lack of Efficacy | 1
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Cholic Acid
Number analyzed (Participants) | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 9 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 24
  More than one race | 0
  Unknown or Not Reported | 22
Region of Enrollment [Number; unit: participants]
  United States | 45
  Argentina | 1
  Canada | 1
  Chile | 1
  Israel | 2
  Italy | 1
  Mexico | 1
  Australia | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Atypical Urinary Bile Acid Excretion by FAB-MS (Fast-Atom-Bombardment Ionization-Mass Spectrometry)
Description: The level of atypical urinary bile acid secretion was scored using a scale of: 0, normal; 1, slight; 2, significant; or 3, marked. A Cochran-Mantel-Haenszel (CMH) test with modified ridit scoring was used to compare the difference between the score at baseline and the worst post-baseline score during treatment with cholic acid in this single-arm trial.
Time Frame: At baseline, then every 12 months for an average of 3.5 years
Population: Patients with values
Measure: Count of Participants; unit: Participants
Arm/Group | Cholic Acid
Number analyzed (Participants) | 51
Participants
  Baseline score: normal | 25
  Baseline score: slight | 6
  Baseline score: significant | 10
  Baseline score: marked | 10
  Worst-post-BL score: normal | 25
  Worst-post-BL score: slight | 11
  Worst-post-BL score: significant | 6
  Worst-post-BL score: marked | 9

2. Secondary Outcome: Evaluation of Serum Transaminases: ALT
Description: Changes in ALT were evaluated in terms of elevations above the upper limit of normal (ULN) and were categorized as: <ULN; ≥1 ULN but <2 ULN; ≥2 ULN but <3 ULN; and ≥3x ULN. Changes from baseline to the worst post-baseline value during treatment with cholic acid in this single-arm trial were presented.
Time Frame: At baseline, then every 12 months for an average of 3.5 years
Population: Patients with values
Measure: Count of Participants; unit: Participants
Arm/Group | Cholic Acid
Number analyzed (Participants) | 48
Participants
  Baseline: ALT<ULN | 27
  Baseline: ULN<=ALT<2 ULN | 9
  Baseline: 2 ULN<=ALT<3 ULN | 7
  Baseline: ALT>=3 ULN | 5
  Worst-post-BL value: ALT<ULN | 20
  Worst-post-BL value: ULN<=ALT<2 ULN | 15
  Worst-post-BL value: 2 ULN<=ALT<3 ULN | 9
  Worst-post-BL value: ALT>=3 ULN | 4

3. Secondary Outcome: Evaluation of Serum Transaminases: AST
Description: Changes in AST were evaluated in terms of elevations above the upper limit of normal (ULN) and were categorized as: <ULN; ≥1 ULN but <2 ULN; ≥2 ULN but <3 ULN; and ≥3x ULN. Changes from baseline to the worst post-baseline value during treatment with cholic acid in this single-arm trial were presented.
Time Frame: At baseline, then every 12 months for an average of 3.5 years
Population: Patients with values
Measure: Count of Participants; unit: Participants
Arm/Group | Cholic Acid
Number analyzed (Participants) | 47
Participants
  Baseline: AST<ULN | 17
  Baseline: ULN<=AST<2 ULN | 17
  Baseline: 2 ULN<=AST<3 ULN | 5
  Baseline: AST<=3 ULN | 8
  Worst-post-BL value: AST<ULN | 15
  Worst-post-BL value: ULN<=AST<2 ULN | 17
  Worst-post-BL value: 2 ULN<=AST<3 ULN | 6
  Worst-post-BL value: AST<=3 ULN | 9

4. Secondary Outcome: Clinical Laboratory Results: Bilirubin
Description: Changes from baseline to the worst post-baseline value during treatment with cholic acid in this single-arm trial for bilirubin. Changes from baseline to the worst post-baseline value during treatment with cholic acid in this single-arm trial were presented in terms of descriptive statistics.
Time Frame: At baseline, then every 12 months for an average of 3.5 years
Population: Patients with values
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Cholic Acid
Number analyzed (Participants) | 48
mg/dL
  Baseline | 3.678 (1.1427)
  Worst-post-BL value | 3.785 (1.1464)

5. Secondary Outcome: Clinical Laboratory Results: Gamma Glutamyl Transferase (GGT)
Description: Changes from baseline to the worst post-baseline value during treatment with cholic acid in this single-arm trial for GGT. Changes from baseline to the worst post-baseline value during treatment with cholic acid in this single-arm trial were presented in terms of descriptive statistics.
Time Frame: At baseline, then every 12 months for an average of 3.5 years
Population: Patients with values
Measure: Mean (Standard Error); unit: U/L
Arm/Group | Cholic Acid
Number analyzed (Participants) | 42
U/L
  Baseline | 38.8 (7.13)
  Worst-post-BL value | 16.4 (8.28)

6. Secondary Outcome: Clinical Laboratory Results: Alkaline Phosphatase
Description: Changes from baseline to the worst post-baseline value during treatment with cholic acid in this single-arm trial for alkaline phosphatase. Changes from baseline to the worst post-baseline value during treatment with cholic acid in this single-arm trial were presented in terms of descriptive statistics.
Time Frame: At baseline, then every 12 months for an average of 3.5 years
Population: Patients with values
Measure: Mean (Standard Error); unit: U/L
Arm/Group | Cholic Acid
Number analyzed (Participants) | 47
U/L
  Baseline | 293.7 (30.30)
  Worst-post-BL value | 39.6 (17.71)

7. Secondary Outcome: Clinical Laboratory Results: Prothrombin Time
Description: Changes from baseline to the worst post-baseline value during treatment with cholic acid in this single-arm trial for prothrombin time. Changes from baseline to the worst post-baseline value during treatment with cholic acid in this single-arm trial were presented in terms of descriptive statistics.
Time Frame: At baseline, then every 12 months for an average of 3.5 years
Population: Patients with values
Measure: Mean (Standard Error); unit: sec
Arm/Group | Cholic Acid
Number analyzed (Participants) | 46
sec
  Baseline | 17.977 (2.1338)
  Worst-post-BL value | 1.045 (2.1442)

8. Secondary Outcome: Physical Examinations: Height
Description: Changes in height percentiles from baseline to the worst post-baseline value during treatment with cholic acid in this single-arm trial.
Time Frame: At baseline, then every 12 months for an average of 3.5 years
Population: Patients with values
Measure: Mean (Standard Error); unit: Height percentiles
Arm/Group | Cholic Acid
Number analyzed (Participants) | 41
Height percentiles
  Baseline | 26.767 (4.4448)
  Worst-post-BL value | 25.540 (4.1064)

9. Secondary Outcome: Physical Examinations: Body Weight
Description: Changes in body weight percentiles from baseline to the worst post-baseline value during treatment with cholic acid in this single-arm trial.
Time Frame: At baseline, then every 12 months for an average of 3.5 years
Population: Patients with values
Measure: Mean (Standard Error); unit: Body weight percentiles
Arm/Group | Cholic Acid
Number analyzed (Participants) | 48
Body weight percentiles
  Baseline | 38.030 (5.2853)
  Worst-post-BL value | 33.227 (4.9842)

10. Secondary Outcome: Incidence of Adverse Events
Description: Number (%) of patients with any AE
Time Frame: At baseline, then every 12 months for an average of 3.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cholic Acid
Number analyzed (Participants) | 53
Participants | 44

ADVERSE EVENTS:
Time Frame: Subjects underwent assessments at baseline and every 12 months or when clinically indicated. Treatment with cholic acid will continue throughout a subject's lifetime. CAC-002-01 study reports data collected from 1 January 2010 until study completion on 31 July 2016, approximately 6.5 years.
Arm/Group | Cholic Acid
All-Cause Mortality (participants affected / at risk) | 6/53
Serious Adverse Events (participants affected / at risk) | 19/53
Other Adverse Events (participants affected / at risk) | 21/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cholic Acid (N=53)
Coagulopathy (Blood and lymphatic system disorders) | 3 (3)
Bradykardia (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Disease progression (General disorders) | 5 (6)
Pyrexia (General disorders) | 1 (1)
Hepatic artery thrombosis (Hepatobiliary disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (2)
Bacteraemia (Infections and infestations) | 1 (1)
Ear infection (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 3 (3)
Sepsis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Encephalopathy (Nervous system disorders) | 2 (2)
Mental impairment (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Adenoidectomy (Surgical and medical procedures) | 1 (1)
Orchidopexy (Surgical and medical procedures) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cholic Acid (N=53)
Abdominal pain (Gastrointestinal disorders) | 6 (8)
Diarrhoea (Gastrointestinal disorders) | 6 (7)
Nasopharyngitis (Infections and infestations) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 8 (8)
Hepatic enzyme increased (Investigations) | 4 (6)
Vitamin D decreased (Investigations) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No